CLINICAL TRIAL: NCT00535158
Title: Vitamin D and Muscle Strength in the Dialysis Population
Brief Title: Vitamin D 2 to Dialysis Patients
Acronym: D2D
Status: Terminated | Type: Observational
Why Stopped: Because of departure of study personnel and lack of funding
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ajay K. Singh, Physician, Brigham and Women's Hospital
Other Study IDs: 2007p-000613
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Kidney Disease; Muscle Weakness; Pain; Fractures, Bone
Keywords: Chronic Kidney disease; Dialysis; Vitamin D; Chronic kidney disease is associated with impaired muscle strength, pain and fractures.
MeSH Terms: conditions — Kidney Diseases; Muscle Weakness; Pain; Fractures, Bone; Renal Insufficiency, Chronic | interventions — Ergocalciferols

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ergocalciferol (Vitamin D 2) — 50,000units once weekly for 8 weeks then every other week for 4 weeks

SUMMARY:
Vitamin D is necessary for healthy bones. Vitamin D is made in our skin when we are exposed to sunlight, but it is also found in foods that we eat and in vitamin pills. Low levels of vitamin D are common in many groups of people, because we do not get enough sun during the winter and because we eat few foods that have vitamin D in them. Some foods with vitamin D are salmon, mackerel, tuna, and fortified milk, which has had vitamin D added to it.

We know that nearly all kidney disease patients on dialysis do not have enough vitamin D in their bodies. We believe this condition can cause muscle weakness, leading to falls and broken bones. These are common problems for patients who are receiving dialysis. For example, dialysis patients have a much higher risk of hip fractures (broken hips). However, no formal research has been done on patients with low vitamin D levels receiving dialysis, to see if they actually have muscle weakness and related problems.

There are two goals of this study. First, we want to see if patients on dialysis who have low vitamin D levels are actually at risk for muscle weakness, muscle pain, and broken bones. We also want to find out if giving vitamin D pills to these patients will result in better muscle strength, less muscle pain, and fewer falls.

In this study, we will compare vitamin D to placebo. Placebo capsules look exactly like vitamin D capsules but contain no active ingredients. We use placebos in research studies to be sure that the study results are due to the study drug and not to other reasons.

DETAILED DESCRIPTION:
Inclusion criteria:

Age ³ 18, CKD on hemodialysis, men and women, hemoglobin ³ 9g/dl, albumin ³ 3.0g/dl, no recent (in the last three months) admissions to the hospital, ability to walk ten feet with or without a walking aid.

Exclusion criteria:

Subjects who are pregnant or lactating; subjects with history of kidney stones, malabsorption syndromes, tertiary hyperparathyroidism defined by a parathyroid hormone of >500pg/ml, current use of corticosteroids, non-ambulatory subjects (for example paraplegic subjects), serious fracture in the last three months, and corrected calcium levels of 10.5 mg/dl or greater.

ELIGIBILITY:
Inclusion criteria:

* Age ³ 18
* CKD on hemodialysis
* Men and women
* Hemoglobin ³ 9g/dl, albumin ³ 3.0g/dl,
* No recent (in the last three months) admissions to the hospital
* Ability to walk ten feet with or without a walking aid.

Exclusion criteria:

* Subjects who are pregnant or lactating
* Subjects with history of kidney stones
* Malabsorption syndromes
* Tertiary hyperparathyroidism defined by a parathyroid hormone of >500pg/ml, current use of corticosteroids
* Non-ambulatory subjects (for example paraplegic subjects)
* Serious fracture in the last three months, and
* Corrected calcium levels of 10.5 mg/dl or greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-01 (Actual)

PRIMARY OUTCOMES:
Vitamin D 2 levels of Dialysis Patients | 1 year

SECONDARY OUTCOMES:
Muscle strength | 1 year
  timed up and go test and dynamometry of four different muscle groups

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Singh, M.D., Principal Investigator — Brigham and Womens Hospital